CLINICAL TRIAL: NCT02281305
Title: Imaging of Inflammation in the Postischemic Myocardium: Effect of Anti-inflammatory Treatment With Colchicine
Brief Title: Post-MI PET Scan Imaging of Inflammation
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: G.Gennimatas General Hospital (Other)
Collaborators: Academy of Athens (Other)
Responsible Party: Principal Investigator, Spyridon Deftereos, Director, Cardiac Catheterization Department, G.Gennimatas General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 22977 / 29-08-2014
Record Dates: First submitted 2014-10-30; First posted 2014-11-03 (Estimated); Last update posted 2014-11-03 (Estimated); Status verified 2014-10

CONDITIONS: Acute Myocardial Infarction
MeSH Terms: interventions — Colchicine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Colchicine Active treatment group (Experimental): Drug: Colchicine 2 mg loading dose; 0.5 mg bid for 5 days
  Interventions: Drug: Colchicine
- Control group (Placebo Comparator): Drug: Placebo

INTERVENTIONS:
Drug: Colchicine
  Arms: Colchicine Active treatment group

SUMMARY:
Restoring the patency of the coronary vessels and providing the ischemic myocardium with reperfused blood can cause additional tissue damage. A key element of ischemia and reperfusion (I/R) injury and major determinant of the evolution of damage in the affected myocardium is the inflammatory response. The main objective of the study is to evaluate the efficacy of colchicine in reducing I/R injury by effectively modulating the inflammatory response in the reperfused myocardium.

ELIGIBILITY:
Inclusion Criteria:

* The study will enroll patients 18 years old or older
* Who presented to the hospital within twelve (12) hours of the onset of chest pain -Who had ST segment elevation > 1 mm in two contiguous limb leads or ST segment elevation > 2 mm in two consecutive precordial leads or new onset of left bundle branch block (LBBB) in a twelve lead electrocardiogram and for whom the decision was made to be taken to the cath lab to perform angioplasty of the coronary vessels.

Exclusion Criteria:

* Excluded patients:

  * with age > 80 years old
  * with active inflammatory diseases, infectious diseases or known malignancy
  * under treatment with corticosteroids, anti-inflammatory agents or disease modifying agents
  * with known hypersensitivity-allergy to colchicine
  * under chronic treatment with colchicine
  * with severe renal failure (eGFR < 30 ml/min/1.73 m2)
  * with hepatic failure (Child - Pugh class B or C)
  * presented with cardiac arrest
  * presented with ventricular fibrillation
  * presented with cardiogenic shock
  * with stent thrombosis
  * with angina within 48 hours before infarction
  * with previous myocardial infarction in the affected territory
  * with occlusion of the left main or left circumflex coronary or the right coronary artery or with evidence of coronary collaterals to the region at risk on initial coronary angiography (at the time of admission)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2014-10; Primary Completion 2015-04 (Estimated)

PRIMARY OUTCOMES:
Degree of inflammation of the involved myocardium as assessed by the PET scan | 5 days post-MI

CONTACTS AND LOCATIONS:
Overall Officials: Constantinos Anagnostopoulos, MD, Principal Investigator — Biomedical Research Foundation of Academy of Athens; Christos Angelidis, MD, Principal Investigator — Athens General Hospital "G. Gennimatas"
Locations (1):
- Athens General Hospital "G. Gennimatas", Athens, Attica, Greece